CLINICAL TRIAL: NCT05729516
Title: The Hope App: An Immersive Telehealth Solution for Older Adults With Diabetes
Brief Title: The Hope App Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: See Yourself Health LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/06/30
Record Dates: First submitted 2022-12-22; First posted 2023-02-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: older adults; telehealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a wait-list control study design. Participants are assigned to one of two groups at random (intervention and wait list) for 6 months. After 6 months, participants in the wait list group are able to receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment Group (ITG) (Experimental): ITG participants receive access to the Hope App, a newly designed immersive learning and telehealth application designed to deliver engaging diabetes care and self-management education and support for older adults with diabetes.
  ITG participants also complete data collection (surveys and HbA1c measurements) at baseline, 3 months after baseline, and 6 months after baseline.
  Interventions: Behavioral: Hope App immersive learning and telehealth platform
- Wait List Control (WLC) (No Intervention): WLC participants receive care as usual for 6 months. They will complete data collection (surveys and HbA1c measurements) at baseline, 3 months after baseline, and 6 months after baseline.
  After 6 months, WLC participants will gain access to the Hope App and receive diabetes programming and health coaching for the remaining 6 months.

INTERVENTIONS:
Behavioral: Hope App immersive learning and telehealth platform — As part of the Hope App intervention, participants attend 10 skills sessions related to diabetes self-management. ITG participants will also receive monthly health coaching calls. After 6 months of active participation, participants enter a maintenance period, during which programming concludes but continued access to the program materials remains.
  Arms: Immediate Treatment Group (ITG)

SUMMARY:
This research study will test how a computer program (called the Hope App) teaches diabetes care skills for older adults with diabetes. The study will compare those who receive diabetes education (10 educational modules and monthly health coaching) through the research program with those who receive care as usual.

DETAILED DESCRIPTION:
The Hope App offers a simple, high-impact, engaging, and immersive telehealth experience with the potential to become a ubiquitous diabetes management tool to transform diabetes patients into high performing drivers of their own care.

The research team aims to scale the platform, develop features that are important to aging adults, and run a clinical trial to validate the Hope App's health benefits.

* Specific Aim 1: Develop the Hope App's state-of-the-art immersive patient engagement experience with automated onboarding, social networking and gamified DSME/S features to support long-term patient retention. In doing so, usability testing will be performed to ensure patient-facing features on the platform and patient-facing content and curriculum materials are functioning and well received by participants.
* Specific Aim 2: Develop the Hope App's predictive analytic capabilities for population health management.
* Specific Aim 3: Conduct a clinical validation trial of the Hope App intervention on six-month clinical outcomes (Hemoglobin A1c), patient reported outcomes (diabetes distress) and engagement outcomes (patient retention, adherence to self-care behaviors).

The research team intends to deliver a scalable Hope App platform with a usable patient engagement portal designed for older adults and achieve decreases in blood glucose levels (HbA1c) and depressive burden, and sustained patient engagement.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years and above
* diagnosis of type 2 diabetes
* English-speaking
* baseline blood sugar value (HbA1c) of 7.5%
* Internet access

Exclusion Criteria:

* aged less than 65 years
* non English-speaking
* unable to provide informed consent
* diagnosis of type 1 diabetes
* unable to use a computer or mobile device
* medical condition for which participation is contraindicated (dialysis, pregnancy, use of insulin pump)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
change in glycemic control | baseline and 6 months
  change in HbA1c values recorded from point-of-care tests or in the electronic health record at visits.
  A mean change of 0.5% will be the a priori determined clinically meaningful minimum improvement from baseline to 6 months.

SECONDARY OUTCOMES:
changes in self-reported diabetes distress | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in diabetes distress scale
self-reported weight change | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported weight change in pounds
changes in participant engagement | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  proportion of utilization metrics met (frequency of use, feature interactions)
changes in self-management adherence | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in the 11-item Summary of Diabetes Self-Care Activities Assessment. The first 10 items are summed to a total score and averaged to 5 scale scores; the scales are General Diet, Specific Diet, Exercise, Blood-Glucose Testing, and Foot Care. Mean number of days will be assessed for self-management behaviors. The 11th question assess smoking status (yes(1), no(0)).
changes in medication adherence scale | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in the Medication Adherence Report Scale (MARS-5). There is also a 10-item version. The 5-item version asks respondents to rate the frequency with which the five different medication-taking behaviors occur, scoring each item on a five-point scale (5 = never to 1 = very often), with higher scores indicating higher levels of adherence to medication.
changes in depressive burden symptoms | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in Patient Health Questionnaire (PHQ)-9. PHQ-9 total score over nine items ranges from 0-24, with higher scores indicative of greater depressive symptom burden.
changes in general anxiety symptoms | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in General Anxiety Disorder (GAD)-7 questionnaire. GAD-7 total score over seven items ranges from 0-21, with higher scores indicative of increased symptoms of anxiety.
changes in coping skills | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes to Brief Resilient Coping Scale. The total score over 4 items ranges from 4-20, with higher scores indicative of high resilient coping.
changes in perceived support from healthcare providers | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in Healthcare Climate Questionnaire
changes in perceived competence | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in Perceived Competence in Diabetes Scale. There are 4-items on a Likert scale from 1-7 with higher scores representing a higher degree to which people with diabetes feel they can self-manage their diabetes. The mean score is used as a summary score.
changes in perceived diabetes self-efficacy | baseline to 3 months; 3 months to 6 months; baseline to 6 months
  self-reported changes in diabetes self-efficacy scale. There are 8 items on a Likert scale from 1 to 10. The score for the scale is the mean of the eight items. Higher number is indicative of higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mitchell, MD, MS, Principal Investigator — See Yourself Health LLC
Locations (1):
- See Yourself Health, Beverly, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No